CLINICAL TRIAL: NCT04776304
Title: Evaluation of Quantitative EEG During Art Therapy in Service Members with Co-Morbid Traumatic Brain Injury & Posttraumatic Stress Symptoms
Brief Title: Art Therapy QEEG Study for Service Members with a Traumatic Brain Injury and Posttraumatic Stress Symptoms
Acronym: ArtTherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: National Intrepid Center of Excellence (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2020-0279
Record Dates: First submitted 2020-04-08; First posted 2021-03-01 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Post-Traumatic Headache; PTSD; TBI; TBI (Traumatic Brain Injury); MTBI - Mild Traumatic Brain Injury; Posttraumatic Stress Disorder; Posttraumatic Stress Disorder, Delayed Onset; Sleep Disturbance; Nightmare; Nightmares, REM-Sleep Type; Headache; Irritable Mood; Anger; Eating Disorders; Combat and Operational Stress Reaction; Combat Stress Disorders; Military Operations; Military Activity; Military Family
MeSH Terms: conditions — Post-Traumatic Headache; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Brain Concussion; Parasomnias; Headache; Feeding and Eating Disorders; Combat Disorders | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: This is both interventional, meaning SMs receive art therapy, and analytical, to understand qEEG outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- qEEG Art Therapy (Other): Participants will receive art therapy while a noninvasive, mobile qEEG measures brain activity. There is no comparison as this is an exploratory pilot study.
  Interventions: Behavioral: Art Therapy

INTERVENTIONS:
Behavioral: Art Therapy — This is a pilot study in which every participant receives the art therapy intervention arm. There are no waitlist or control arms. Art therapy is one promising intervention that helps service members (SMs) develop a "visual voice," using imagery, symbolism, and metaphor to externalize emotions and experiences that they may not be able to express in words. The standardized, integrative mental health and human services approach of the art therapy program at the NICoE utilizes a mask-making directive to explore thoughts, feelings, and experiences of combat and self-understanding. This process is especially relevant to SMs with PTS symptoms who often remember their trauma as an incoherent, fragmented memory that is often predominantly sensory in nature. NICoE researchers have provided preliminary evidence suggesting associations between recurring art themes represented within the masks and individual BH symptoms.

SUMMARY:
Service members and/or recently separated veterans with post traumatic stress symptoms and mild traumatic brain injury may participate in 8 sessions including 2 sessions including interviews and questionnaires as well as 6 sessions of art therapy. In the art therapy, participants will be provided with a blank paper mache mask template and invited to alter the mask however they wish using a variety of art materials. The therapist will use the art-making process and culminating product to aid in self-reflection, reframe negative thoughts and feelings, and work through traumatic content. Prior to the session start participants will get set up with a mobile qEEG (worn like a hat and backpack). The qEEG will measure brain activity in a non-invasive way throughout the art therapy session to improve understanding of brain activity during the art therapy process.

DETAILED DESCRIPTION:
This is a pilot, interventional clinical trial in which all 9 service members with comorbid PTSD and mTBI participate in 8 sessions (1 baseline session of interviews and questionnaires, 6 sessions of art therapy, and 1 final session of interviews and questionnaires). Participants must have significant posttraumatic stress symptoms and a history of mild traumatic brain injury. Target enrollment is 9 active duty service members or recently separated veterans, aged 18-64 with no prior art therapy exposure, at the NICoE at Walter Reed National Military Medical Center in Bethesda, MD.

Background: Posttraumatic stress disorder (PTSD) and mild traumatic brain injury (mTBI) are persistent and frequently comorbid complications of combat that remain a challenge to healthcare providers. In these complex cases, traditional treatments often fail to provide complete relief from symptoms associated with posttraumatic stress (PTS), anxiety, and depression, leading the military healthcare system to look towards complementary and integrative treatments. Art therapy is one promising intervention that helps service members (SMs) develop a "visual voice," using imagery, symbolism, and metaphor to externalize emotions and experiences that they may not be able to express in words. The standardized, integrative mental health and human services approach of the art therapy program at the NICoE utilizes a mask-making directive to explore thoughts, feelings, and experiences of combat and self-understanding. This process is especially relevant to SMs with PTS symptoms who often remember their trauma as an incoherent, fragmented memory that is often predominantly sensory in nature. NICoE researchers have provided preliminary evidence suggesting associations between recurring art themes represented within the masks and individual BH symptoms; yet, the neurobiological mechanisms underlying this therapeutic technique remain obscure. To date, there have been few studies using neuroimaging techniques to investigate brain network changes during art creation. Studies have utilized electroencephalography (EEG) and functional near infrared spectroscopy (fNIRS) during art creation but not within the context of art therapy. Mobile, quantitative EEG allows for real time data capture that could minimize interference of neuroimaging during the therapeutic process and provide insight into the neurological mechanisms underlying art therapy.

Study design and procedures: Participants will be provided with a blank paper mache mask template and invited to alter the mask however they wish using a variety of art materials. The therapist will use the art-making process and culminating product to aid in self-reflection, reframe negative thoughts and feelings, and work through traumatic content. Prior to the session start participants will get set up with the mobile qEEG. The qEEG will be segmented into a pre-art therapy session resting state, prompt-specific tasks during the art therapy session, and a post-art therapy session resting state.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service member or recently separated veteran (within the past 5 years)
* DEERs eligible
* Significant posttraumatic stress symptoms
* History of mild traumatic brain injury
* Aged 18-64

Exclusion Criteria:

* Previous art therapy exposure
* Moderate, severe, or penetrating TBI history
* History of a psychotic disorder, bipolar disorder, or active suicidal or homicidal ideation
* Unable to provide informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is an analysis of qEEG session data. | during the intervention Session 1 (Week 2)
  The primary outcome measure is an analysis of qEEG session data, which will include regional and global power across the following frequency bands: delta (1-4 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (13- 30 Hz), and gamma (>30 Hz); global interhemispheric coherence; and regional coherence between pairs of sensor locations. Global/regional power (units: micro-Volts-squared per Hz (uV2/Hz) Interhemispheric coherence (units coherence) Regional coherence (units coherence)
The primary outcome measure is an analysis of qEEG session data. | during the intervention Session 2 (Week 3)
  The primary outcome measure is an analysis of qEEG session data, which will include regional and global power across the following frequency bands: delta (1-4 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (13- 30 Hz), and gamma (>30 Hz); global interhemispheric coherence; and regional coherence between pairs of sensor locations. Global/regional power (units: micro-Volts-squared per Hz (uV2/Hz) Interhemispheric coherence (units coherence) Regional coherence (units coherence)
The primary outcome measure is an analysis of qEEG session data. | during the intervention Session 3 (Week 4)
  The primary outcome measure is an analysis of qEEG session data, which will include regional and global power across the following frequency bands: delta (1-4 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (13- 30 Hz), and gamma (>30 Hz); global interhemispheric coherence; and regional coherence between pairs of sensor locations.Global/regional power (units: micro-Volts-squared per Hz (uV2/Hz) Interhemispheric coherence (units coherence) Regional coherence (units coherence)
The primary outcome measure is an analysis of qEEG session data. | during the intervention Session 4 (Week 5)
  The primary outcome measure is an analysis of qEEG session data, which will include regional and global power across the following frequency bands: delta (1-4 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (13- 30 Hz), and gamma (>30 Hz); global interhemispheric coherence; and regional coherence between pairs of sensor locations. Global/regional power (units: micro-Volts-squared per Hz (uV2/Hz) Interhemispheric coherence (units coherence) Regional coherence (units coherence)
The primary outcome measure is an analysis of qEEG session data. | during the intervention Session 5 (Week 6)
  The primary outcome measure is an analysis of qEEG session data, which will include regional and global power across the following frequency bands: delta (1-4 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (13- 30 Hz), and gamma (>30 Hz); global interhemispheric coherence; and regional coherence between pairs of sensor locations. Global/regional power (units: micro-Volts-squared per Hz (uV2/Hz) Interhemispheric coherence (units coherence) Regional coherence (units coherence)
The primary outcome measure is an analysis of qEEG session data. | during the intervention Session 6 (Week 7)
  The primary outcome measure is an analysis of qEEG session data, which will include regional and global power across the following frequency bands: delta (1-4 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (13- 30 Hz), and gamma (>30 Hz); global interhemispheric coherence; and regional coherence between pairs of sensor locations. Global/regional power (units: micro-Volts-squared per Hz (uV2/Hz) Interhemispheric coherence (units coherence) Regional coherence (units coherence)

SECONDARY OUTCOMES:
CAPS-5 | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Clinician-Administered PTSD Scale for DSM-5
TAS-20 | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  The Toronto Alexithymia Scale
AIQ | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Aspects of Identity Questionnaire
PCL-5 | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Post Traumatic Stress Symptom Questionnaire
GAD-7 | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  General Anxiety Disorder Questionnaire
PHQ-9 | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Patient Health Questionnaire for depression symptoms
PHQ-15 | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Patient Health Questionnaire for somatic symptoms
NSI | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Neurological Symptom Inventory
PGIC | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  General Impression of Change
SUD Scores | baseline (pre-intervention) and immediately after the intervention; within a period of 8 weeks
  Subjective Units of Distress

CONTACTS AND LOCATIONS:
Locations (1):
- National Intrepid Center of Excellence at Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No